CLINICAL TRIAL: NCT04714164
Title: Feasibility of Delivering Group Cognitive Behavioral Therapy for Older Adults With Depression and Anxiety by Telehealth
Brief Title: Cognitive Behavioral Therapy Group for Older Adults Delivered by Telethealth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We had difficulty with participation in the study for our initial Zoom CBT group.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29243
Record Dates: First submitted 2021-01-07; First posted 2021-01-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder

STUDY DESIGN:
Intervention Model Description: Feasibility and acceptability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teletherapy Group CBT participants (Experimental): Patients over the age of 65 with either a Major Depressive Disorder or Generalized Anxiety Disorder who will be participating in a Group CBT delivered by Teletherapy
  Interventions: Behavioral: Group Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — Therapy will be delivered weekly for 8 weeks by Zoom.

SUMMARY:
The present aim of the study is to to adapt an established, manualized enhanced Group CBT (CBT-E) for seniors to a telehealth format, which will allow us to offer the group virtually during the COVID-19 pandemic.

DETAILED DESCRIPTION:
The goal of this project is to adapt an established, manualized enhanced Group CBT (CBT-E) for seniors to a telemedicine format. Currently the Geriatric Psychiatry service associated with the Nova Scotia Health Authority offer two CBT-E groups every year. They are usually facilitated by psychiatry residents, under the supervision of a staff psychiatrist. Due to the risk of COVID-19, we will not be holding in-person groups this year. Instead we will offer the group in a smaller, telemedicine format. For this project, we will change the group structure and activities to allow it's delivery in a virtual format. This study will assess feasibility, tolerability of the telehealth format by using the System Usability Scale and Group Satisfaction Survey. It will also assess response to online therapy buy using pre- and post-group questionnaires including the Beck Depression Inventory, Beck Anxiety Inventory and Perceived Quality of Life Questionnaire. Paired t-tests will be used to analyse the data and determine whether there has been an improvement in participant's symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* People over the age of 65
* Diagnosis of either or both Major Depressive Disorder (MDD) of mild or moderate severity and an anxiety disorder, including generalized anxiety disorder, social anxiety disorder or panic disorder.

Exclusion Criteria:

* Patients with psychosis
* Patients with dementia
* Patient with severe Major Depressive Disorder or Anxiety Disorder
* Patients with antisocial or borderline personality disorder
* Patients with acute suicidal ideation.
* Older adults who do not have access to the technology required for group; computer, phone or tablet with a webcam and access to Internet

These are also exclusion criteria for the CBT group outside of the study. People younger than 65 are also excluded from the group because it is offered to older adults only.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of Telehealth CBT group for older adults | This will be completed at the end of the 8 week Telehealth CBT group.
  This will be assessed by a questionnaire: System Usability Scale.
Acceptability of Telehealth CBT group for older adults | This will be completed at the end of the 8 week Telehealth CBT group.
  This will be measured by a questionnaire administered to participants titled Satisfaction Survey.
Attrition to the Telehealth CBT group for older adults | 8 weeks
  Attendance will be noted by group facilitators at each group session

SECONDARY OUTCOMES:
Effect size between pre-group and post-group questionnaires (anxiety) | Scales will be administered at baseline and at the end of the 8 weeks of group therapy.
  The following scale will be administered before and after completing the group to determine if there is any change in the result: Beck Anxiety Inventory.
Effect size between pre-group and post-group questionnaires (depression) | Scales will be administered at baseline and at the end of the 8 weeks of group therapy.
  The following scale will be administered before and after completing the group to determine if there is any change in the result: Beck Depression Inventory.
Effect size between pre-group and post-group questionnaires (perceived quality of life) | Scales will be administered at baseline and at the end of the 8 weeks of group therapy.
  The following scale will be administered before and after completing the group to determine if there is any change in the result: Perceived Quality of Life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Boudreau, MD, Principal Investigator — NSHA
Locations (1):
- Abbie J Lane Memorial Building - QEII, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hendriks GJ, Oude Voshaar RC, Keijsers GP, Hoogduin CA, van Balkom AJ. Cognitive-behavioural therapy for late-life anxiety disorders: a systematic review and meta-analysis. Acta Psychiatr Scand. 2008 Jun;117(6):403-11. doi: 10.1111/j.1600-0447.2008.01190.x. PMID 18479316
- [Background] Tavares LR, Barbosa MR. Efficacy of group psychotherapy for geriatric depression: A systematic review. Arch Gerontol Geriatr. 2018 Sep-Oct;78:71-80. doi: 10.1016/j.archger.2018.06.001. Epub 2018 Jun 18. PMID 29933137
- [Background] O'Reilly R, Bishop J, Maddox K, Hutchinson L, Fisman M, Takhar J. Is telepsychiatry equivalent to face-to-face psychiatry? Results from a randomized controlled equivalence trial. Psychiatr Serv. 2007 Jun;58(6):836-43. doi: 10.1176/ps.2007.58.6.836. PMID 17535945
- [Background] Gentry MT, Lapid MI, Rummans TA. Geriatric Telepsychiatry: Systematic Review and Policy Considerations. Am J Geriatr Psychiatry. 2019 Feb;27(2):109-127. doi: 10.1016/j.jagp.2018.10.009. Epub 2018 Oct 30. PMID 30416025
- [Background] Wilson KC, Mottram PG, Vassilas CA. Psychotherapeutic treatments for older depressed people. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD004853. doi: 10.1002/14651858.CD004853.pub2. PMID 18254062
- [Background] Hantke N, Lajoy M, Gould CE, Magwene EM, Sordahl J, Hirst R, O'Hara R. Patient Satisfaction With Geriatric Psychiatry Services via Video Teleconference. Am J Geriatr Psychiatry. 2020 Apr;28(4):491-494. doi: 10.1016/j.jagp.2019.08.020. Epub 2019 Aug 24. PMID 31530457
- [Background] Hubley S, Lynch SB, Schneck C, Thomas M, Shore J. Review of key telepsychiatry outcomes. World J Psychiatry. 2016 Jun 22;6(2):269-82. doi: 10.5498/wjp.v6.i2.269. eCollection 2016 Jun 22. PMID 27354970
- [Background] Baldwin RC, Anderson D, Black S, Evans S, Jones R, Wilson K, Iliffe S; Faculty of Old Age Psychiatry Working Group, Royal College of Psychiatrists. Guideline for the management of late-life depression in primary care. Int J Geriatr Psychiatry. 2003 Sep;18(9):829-38. doi: 10.1002/gps.940. PMID 12949851
- [Background] Apostolo J, Bobrowicz-Campos E, Rodrigues M, Castro I, Cardoso D. The effectiveness of non-pharmacological interventions in older adults with depressive disorders: A systematic review. Int J Nurs Stud. 2016 Jun;58:59-70. doi: 10.1016/j.ijnurstu.2016.02.006. Epub 2016 Feb 17. PMID 27087298
- [Background] Jonsson U, Bertilsson G, Allard P, Gyllensvard H, Soderlund A, Tham A, Andersson G. Psychological Treatment of Depression in People Aged 65 Years and Over: A Systematic Review of Efficacy, Safety, and Cost-Effectiveness. PLoS One. 2016 Aug 18;11(8):e0160859. doi: 10.1371/journal.pone.0160859. eCollection 2016. PMID 27537217
- [Background] Choi NG, Marti CN, Bruce ML, Hegel MT, Wilson NL, Kunik ME. Six-month postintervention depression and disability outcomes of in-home telehealth problem-solving therapy for depressed, low-income homebound older adults. Depress Anxiety. 2014 Aug;31(8):653-61. doi: 10.1002/da.22242. Epub 2014 Feb 5. PMID 24501015
- [Background] Egede LE, Acierno R, Knapp RG, Lejuez C, Hernandez-Tejada M, Payne EH, Frueh BC. Psychotherapy for depression in older veterans via telemedicine: a randomised, open-label, non-inferiority trial. Lancet Psychiatry. 2015 Aug;2(8):693-701. doi: 10.1016/S2215-0366(15)00122-4. Epub 2015 Jul 16. PMID 26249300
- [Background] MacQueen GM, Frey BN, Ismail Z, Jaworska N, Steiner M, Lieshout RJ, Kennedy SH, Lam RW, Milev RV, Parikh SV, Ravindran AV; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 6. Special Populations: Youth, Women, and the Elderly. Can J Psychiatry. 2016 Sep;61(9):588-603. doi: 10.1177/0706743716659276. Epub 2016 Aug 2. PMID 27486149
- See also: Center for Multicultural Mental Health Research 2012 — https://www.multiculturalmentalhealth.ca/en/
- See also: Yalom, I.D., The Theory and Practice of Group Psychotherapy, 5th edition, Basic Books — https://www.basicbooks.com/titles/irvin-d-yalom/the-theory-and-practice-of-group-psychotherapy/9780465012916/
- See also: National Institute for Clinical Excellence. Depression: management of depression in primary and secondary care. NICE 2004. — https://www.nice.org.uk/